CLINICAL TRIAL: NCT05151822
Title: Virtual Reality in Awake Surgery : Pilot Study VIRAS
Acronym: VIRAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC21.0039 (VIRAS)
Record Dates: First submitted 2021-11-08; First posted 2021-12-09 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Surgery
Keywords: Awake surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual reality mask (Experimental): Realization of the following examinations with virtual reality mask :
  * Training session
  * Acceptability of the device before and after surgery
  * Monitoring of the device during surgery
  Interventions: Other: Training session with the virtual reality mask; Other: Monitoring of the device; Other: Acceptability of the device; Other: Patient state of anxiety

INTERVENTIONS:
Other: Training session with the virtual reality mask — Patients will have a training session with the virtual reality mask, the day before surgery. The training consists in the realization, by the patient, of a series of language or neuropsychological tests and evaluation of the acceptability of the device by the patient with Visual Analog Scale (device tolerance from 0 (intolerable) to 10 (completely tolerated)).
Other: Monitoring of the device — In the operating room : installation and per-operative monitoring of the device. If the device was removed, the list of device side effects or surgery-related adverse events that was required discontinuation of the device will be established.
Other: Acceptability of the device — After the surgery: evaluation of the acceptability of the device by the patient with Visual Analog Scale (device tolerance from 0 (intolerable) to 10 (completely tolerated))
Other: Patient state of anxiety — Assessing patient's state of anxiety with the State-Trait Anxiety Inventory (STAI) after surgery.

SUMMARY:
The virtual reality mask is a tool likely to improve the conditions for performing awake surgery:

* by improving tolerance for the patient,
* by improving ergonomics in the operating room.

In order to control the risks as well as possible, the investigators propose to test the equipment on patients who will undergo orthopedic surgery under local anesthesia at the hospital of Brest: the patients operated in orthopedics under local anesthesia are immobile during the procedure. This target population will allow an immersion of the equipment in the operating room, with an awake patient, during a short time (on average 1 hour of intervention) and for a technically light interventional procedure.

ELIGIBILITY:
Inclusion Criteria :

* Major subject
* Consent for the study
* Patients eligible for orthopedic surgery with local anesthetic block
* Estimated duration of the Orthopedic surgery of minimum 1 hour

Exclusion Criteria :

* Age < 18 years, Age > 75 years,
* Known central neurological pathology/cognitive impairment,
* Mini-Mental State examination (MMSe) < 23 if no school certificate, < 27 if school certificate,
* History of vertigo,
* Claustrophobia,
* Visual deficit not compatible with the use of the virtual reality mask,
* Contraindication to surgery,
* Outpatient treatment,
* Refusal or inability to consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Tolerance of minimum 1 hour of the virtual reality mask (realization, by the patient, of a series of of language or neuropsychological tests) | 1 Day
  Study the tolerance of the virtual reality mask on patients in the operating room for orthopedic surgery under loco-regional anesthesia. The mask must be maintained during the testing (minimum 1 hour). The testing consists in the realization, by the patient, of a series of language or neuropsychological tests predefined during the preoperative assessment.

SECONDARY OUTCOMES:
Device-related adverse event | 1 Day
  List of device-related adverse events with Simulator Sickness Questionnaire (SSQ). SSQ quantified virtual reality mask sickness with 16 questions on a self-report basis.
Withdrawal of the device | 1 Day
  List of adverse events that required removal of the device (device side effects or surgery-related adverse events that may require discontinuation of the device)
Device tolerance for the patient | 1 Day
  Visual Analog Scale (VAS) of device tolerance from 0 (intolerable) to 10 (completely tolerated), immediately after the training session and at the end of the procedure.
Device tolerance for the medical staff | 1 Day
  Visual Analog Scale (VAS) of device tolerance from 0 (intolerable) to 10 (completely tolerated), to a representative of each profession present in the operating room during the procedure (anesthetist, surgeon, nurse), at the end of the procedure
Patient state of anxiety | 1 Day
  Assessing patient's state of anxiety with the STAI. The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Higher scores are positively correlated with higher levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Pr SEIZEUR Romuald, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending 15 years following the last visit of the last patient.
Access Criteria: Data access requests will b reviewed be the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.